CLINICAL TRIAL: NCT06670937
Title: Role of BARriers in IgG-Pathogen Interactions at the Mucosal Surface in Human Airways
Acronym: BARRIG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DR240158
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Bronchiectasis Adult
Keywords: induced sputum; IgG
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This study aims at collecting airway mucus from individuals with non cystic fibrosis bronchiectasis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): This is the single arm of this study. Patients with non-CF bronchiectasis will provide 1) an induced sputum sample after inhaling 15 ml of 0.9% NaCl solution and 2) a blood sample.
  Interventions: Other: Induced sputum; Other: Blood sample

INTERVENTIONS:
Other: Induced sputum — Patients will provide 1) an induced sputum sample after inhaling 15 ml of 0.9% NaCl solution
Other: Blood sample — Patients will provide 2) a blood sample.

SUMMARY:
Context. Non cystic fibrosis bronchiectasis (NCFB) is a group of suppurative chronic airway diseases of multiple causes. Bronchiectasis is characterized by an abnormal, irreversible dilatation of the bronchi, airway obstruction, chronic cough, and sputum production. Inhaled polyclonal immunoglobulin G (IgG) is a new therapeutic approach for NCFB. Inhaled IgG is expected to have beneficial effects due to its ability to reduce the range of respiratory pathogens capable of infecting the respiratory tract, decrease the pulmonary load of existing bacterial populations, improve mucociliary clearance by restoring epithelial cell functions, and decrease lung inflammation. Pre-clinical data packages showed that IgG reduced the airway pathogen load and related cell damage after infection in rodents and non-human primates. The aim of this study is collect information on the impact of NFCB airway mucus on the biological barriers to locally delivered IgG.

Study design. Thirty patients with stable NFCB will be recruited. The patients will provide induced sputum samples after inhaling isotonic saline. Induced sputum will be used for 1) identification of colonizing bacteriological, fungal and virological populations and 2) for in vitro pharmacological experiments.

The main outcome is the quantification by whole-cell ELISA of binding to Pseudomonas aeruginosa by a polyclonal IgG in the presence of mucus derived from the sputum of NCFB patients.

Secondary outcomes are (1) the measurement of proteolysis, by Western-Blot, of exogenous polyclonal IgG added in the mucus derived from sputum of NCFB patients. The results will be expressed as a percentage of integrity over the one obtained when the polyclonal IgG is added in saline solution and will be compared with in vitro results; (2) the measurement of mobility by Fluorescence Recovery After Photobleaching (FRAP) of exogenous fluorescently-labelled polyclonal IgG added in the mucus derived from sputum of NCFB patients. The results will include the determination of the t(1/2), mobile and immobile fractions over the one obtained when the polyclonal IgG is added in saline solution and will be compared with in vitro results; (3) impact of microbial airway colonization on IgG binding, proteolysis and Ig mobility. Samples with microbial colonization (either bacterial, viral or fungal) will be compared with uncolonized samples.

This project will help in decision-making in the development of inhaled antibody therapeutics. Specifically, the study will provide information on the capacity of locally applied polyclonal IgG to diffuse through mucus and bind to pathogens.

DETAILED DESCRIPTION:
Since the advent of monoclonal antibody technology, therapeutic antibodies (Ab) have proven successful for the treatment of a variety of diseases. Ab radically changed the management and treatment of fatal diseases, ranging from non-Hodgkin's lymphoma to subtypes of asthma. The success of Ab is based on their high selectivity, predictable toxicity and unique pharmacological profiles, giving them advantages over small molecule drugs. As a result, Ab represents the fastest growing class of biotherapeutics, with five of them among the best-selling drugs in the USA.

Respiratory diseases affect millions of people worldwide; the four most commonly fatal lung diseases (pneumonia, tuberculosis, lung cancer, and chronic obstructive pulmonary disease [COPD]) account for about one in five deaths worldwide in 2030 according to WHO. In addition to premature mortality, respiratory diseases have a dramatic impact on society with respect to disability, healthcare costs, and productivity loss, urging the necessity of new therapeutics. With over 100 molecules under clinical evaluation and a dozen of antibodies (Ab) which have received marketing approval, Ab have a tremendous opportunity to benefit patients with respiratory diseases, including bronchiectasis. Presently, Ab are indicated as alternative or complementary strategies to anti-tumour, anti-inflammatory and anti-infectious agents, in particular to antibiotics. The behaviour of Ab depends on their pharmacodynamics (PD) and pharmacokinetics (PK), which partly depend on their route of administration. Up to now, Ab for respiratory diseases are mainly administered intravenously or subcutaneously, which is not optimal to ensure a therapeutic concentration of the active drug in the lungs while it exposes other organs to the drug.

For the treatment of respiratory diseases, inhalation allows to directly target the respiratory tract. Inhalation aims at delivering drugs topically - as an aerosol - through the nose and/or mouth to its site of action. Inhalation is the gold standard for the delivery of drugs with topical action to treat asthma or COPD. Inhalation provides a better therapeutic index for some drugs, often requires reduced dose as compared to other routes, and is non-invasive, thereby improving treatment adherence and patient comfort. Presently, most (topical) inhaled drugs are small molecules from different classes. Ab are usually full-length IgG, which are large heterodimeric proteins (~150 kDa) that do not diffuse passively across cellular barriers. Currently the majority of Ab for respiratory diseases is delivered by the intravenous route (i.v). The i.v. route may not be optimal for Ab in the context of respiratory disease, since only a small fraction of Ab reaches the lungs/airways after i.v. injection. Inhalation is an attractive and feasible alternative route for the topical delivery of full-length Ab into the lungs. Ab delivered through the airway exhibit therapeutic responses and are mostly retained in the lung with low systemic diffusion. Overall, these findings indicate that inhalation may have the edge over other routes of administration when Ab are intended to operate in the respiratory tract.

Despite the theoretical advantages of topical administration of Ab by inhalation, few of these benefits have yet materialized in the clinics. Presently several Ab are in clinical development by inhalation, but none yet in the clinics. This paucity highlights the complexity of developing inhaled antibodies and points out the persisting hurdles to overcome. A detailed understanding of the pharmacology of inhaled Ab is required to ensure the successful transition from pre-clinical to clinical development. In particular, the deposition of Ab aerosol during respiratory diseases may be modulated by biological barriers, which may limit or prevent aerosolized Ab efficacy. Presently, the events that occur after inhaled Ab has deposited in the airways are incompletely known and require deeper characterization.

Non cystic fibrosis bronchiectasis (NCFB) is a group of suppurative chronic airway diseases of multiple etiologies. Clinically, NFCB is characterized by an abnormal, irreversible dilatation of the bronchi, airway obstruction, chronic cough and increased sputum production. At the pathophysiological level, chronic inflammation, chronic airway bacterial colonization and increased airway mucus production play key roles. Current treatment for microbial colonization and/or acute exacerbations of NFCB mostly relies on high-dose systemic or airway-delivered antibiotics. Low-dose long-term azithromycin is also used often used to reduced airway inflammation, symptoms, and the frequency of acute exacerbations. Since antibiotics may either fail to improve symptoms or drive microbial resistance, there is a need for new treatments to improve pathogen clearance and reduce airway inflammation.

Inhaled polyclonal immunoglobulin G (IgG) is a new therapeutic approach for NCFB. Inhaled IgG is expected to mediate beneficial effects in NCFB due to its ability to reduce the range of respiratory pathogens capable of infecting the respiratory tract, decrease the pulmonary load of existing bacterial populations, improve mucociliary clearance by restoring epithelial cell functions, and decrease lung inflammation. Indeed, pre-clinical data packages showed a reduced pathogen load and related cell damage after infection in rodents and non-human primate. A phase 1 trial in NCFB patients and a chronic toxicology study to enable a phase 2 trial, including daily and prophylactically administration of nebulised IgG over 6 months in NCFB patients, are currently underway (NCT00322556, NCT00168025, NCT00168012, NCT00520494).

In NCFB, airway mucus may act as a barrier to inhaled drugs at the mucosal interface. While normal mucus presents as a thin layer that allows IgG to diffuse efficiently to the underlying tissues, airway mucus in NCFB is present in increased amounts and is abnormally thick. Impairment of mucus amount, structure and fluidity during bronchiectasis may thus limit penetration of inhaled Ab and their therapeutic potential. Patients with NCFB also frequently present with chronic bacterial airway colonization and chronic airway inflammation characterized by increased protease activity. They also often suffer from exacerbations, which are pathogen (notably P. aeruginosa and influenza virus)-driven episodes of increased symptoms that require medical intervention, often including the administration of antibiotics. In the context of excessive inflammation, the amount of proteases overwhelms the neutralizing capacity of endogenous protease inhibitors. This may have a dramatic impact on inhaled Ab metabolism and limit their efficacy. Indeed, previous reports show that IgG proteolysis mediated by neutrophil-derived elastase leads to a decrease of anti-P. aeruginosa phagocytosis and killing. In addition to endogenous enzymes (mainly serine [neutrophil-derived] and cysteine [cathepsin] proteases), bacterial pathogens, like P. aeruginosa, also secrete proteases, which may degrade respiratory-delivered drugs. In addition, pathogens like P. aeruginosa induce mucin expression.

During a first in vitro study, we evaluated the barrier effect of artificial mucus with viscosity in the range of that measured in mucus derived from sputum of patients with respiratory diseases. CEPR observed a significant alteration of the mobility and diffusion of the polyclonal IgG (CSL Behring) exogenously added, dependent on the viscosity of the ASM. Importantly, CEPR also determined a significant reduction in the ability of the polyclonal IgG to bind to P. aeruginosa in the presence of viscous mucus in comparison to fluid mucus.

Study objectives. The main objective is to evaluate the impact of mucus derived from sputum of NCFB patients on the binding of a polyclonal IgG to Pseudomonas aeruginosa. Results obtained with NCFB patient mucus will be compared with results obtained using artificial mucus. Secondary objectives are characterization of 1) exogenous polyclonal IgG mobility and 2) stability in the mucus derived from sputum of NCFB patients. In addition, the impact of microbial airway colonization on IgG 's pharmacodynamics will be explored.

Study design. This is an exploratory, prospective, monocentric, cross-sectional, interventional with minimal risks and constraints study of patients with non-cystic fibrosis bronchiectasis (NCFB) followed by the rare pulmonary diseases centre and Pulmonology department of Tours University Hospital (CHRU Tours). The patients included in the study will continue their usual follow-up. The usual medical management - diagnostic and/or therapeutic - will not be modified by participation in the study apart from an additional microbiological study of sputum as part of the study.

This study will focus on the analysis of the biochemical and biophysical properties of a therapeutic polyclonal IgG preparation in the presence of sputum isolated from NCFB patients, and more specifically on the ability of IgG to recognize a target. Mobility and stability of IgG in airway mucus will also be evaluated. In order to associate PD endpoints - measured at the CEPR - with clinically relevant parameters, sputum collection will be accompanied by documentation, in the mucus and blood, of microbiological (virological and bacteriological analyses) and inflammatory (blood formulation, C-reactive protein) parameters - measured at the CHRU of Tours.

Analyzes in the blood compartment will be carried out using an additional volume of blood taken at the time of the visit, respecting the limits and contraindications (in accordance with the order of April 4, 2018 of article L.1121-1 of the Public health code). The analysis in the airways will be carried out using sputum collected from patients. A single analysis point will be planned for each patient included in the study.

Outcome measures. The main outcome is the quantification of polyclonal IgG binding to Pseudomonas aeruginosa in the presence of mucus derived from sputum of NCFB patients. Binding will be assessed by whole-cell ELISA.

The results will be expressed as a percentage of binding over the one obtained when the polyclonal IgG is added in saline solution and will be compared with artificial mucus preparations in a range of viscosity similar to human airway mucus.

Secondary outcomes are: (1) the measurement of proteolysis, by Western-Blot, of exogenous polyclonal IgG added in the mucus derived from sputum of NCFB patients. The results will be expressed as a percentage of integrity over the one obtained when the polyclonal IgG is added in saline solution and will be compared with in vitro results; (2) the measurement of mobility by FRAP of exogenous fluorescently labelled polyclonal IgG added in the mucus derived from sputum of NCFB patients. The results will include the determination of the t(1/2), mobile and immobile fractions over the one obtained when the polyclonal IgG is added in saline solution and will be compared with in vitro results. This will be done at the CEPR. (3) impact of microbial airway colonization on IgG binding, proteolysis and Ig mobility. Samples with microbial colonization (either bacterial, viral or fungal) will be compared with uncolonized samples.

Selection and recruitment of people suitable for research. Study population includes all patients with an age ≥ 18 years suffering from NCFB and followed by the rare pulmonary diseases centre / Pulmonology department of CHRU Tours (active list comprises 181 patients with idiopathic NFCB on September 2023). These patients routinely attend clinic visit including forced spirometry at least yearly. In this cross-sectional study, patients will be screened based on medical records from the Rares Pulmonary Diseases Center at Tours university hospital (CHRU Bretonneau). In particular, patients will be screened for chronic sputum production. It is estimated that a third of all patients may be eligible for the study. Eligible patients will be offered to participate either at the time of a scheduled visit to the hospital, or by a phone call by a research assistant or research nurse. Patients interested in the study will be provided the information document for further information. When patients give oral consent to participate in the study, they will be invited to come for a visit at the Clinical Investigation Center (CIC Inserm 1415) of the hospital. Patients will then meet an investigator. To be involved, a subject must fulfil all inclusion criteria and no non-onclusion criteria. Consent will be confirmed by the investigator after a meeting with the subject and review of the letter of consent.

Study visit. At inclusion, patient will attend a visit by an investigator to record clinical examination and vital signs, date of latest acute exacerbation, medical history, treatment, and Saint George's respiratory questionnaire (quality of life measure). Description of bronchiectasis from the latest computed tomography scan (CT), severity of lung function impairment defined by the latest spirometry (FEV1), and bronchiectasis severity index, will be validated by a senior pulmonologist.

Clinical data collection.

At inclusion, patient will attend a visit by an investigator to record:

* Medical history
* Current treatment
* Clinical examination and vital signs (blood pressure, heart rate, percutaneous haemoglobin saturation-SPO2 while breathing room air)
* mMRC dyspnea scale
* Description of bronchiectasis severity from the latest CT, using the Bronchiectasis Radiologically Indexed CT Score (BRICS) and the number of lobes involved 19
* Severity of airflow impairment (forced expiratory in 1 second-FEV1) from the latest spirometry. FEV1 is expressed as percent of the predicted value using GLI2012 reference equations
* Date of latest acute exacerbation (defined as increased respiratory symptoms lasting >48h and a new antibiotic prescription)
* Number and date of severe exacerbations requiring hospitalization
* Number of acute exacerbations requiring antibiotic therapy in the past year
* Saint George's respiratory questionnaire (quality of life measure)
* History of airway colonization by Pseudomonas or other bacteria

Blood and inhaled sputum sample collection. Following the medical consultation 3x5 mL venous blood will be drawn by a CIC nurse for haematological and biochemical analyses. 1 tube will be used for immunological analysis made at the CEPR.

Following blood collection, subjects will receive a 0.9% NaCl aerosol if SPO2 while breathing room air is ≥94%, and induced sputum samples will be collected. The key steps of aerosol delivery and sputum collection are :

* The patient rinses his/her mouth with drinking water (to reduce contamination of the sample with saliva)
* The patient blows his/her nose (to reduce contamination of the sample with upper airway mucus)
* Begin nebulization of 15 mL 0.9% NaCl delivered via a pneumatic nebuliser (6L/min air)
* During and immediately after the NaCl aerosol, the subject is encouraged to expectorate into a 50 mL sampling tube at least 3 times (5, 10, 15 minutes).

Sample analysis. Immediately following collection, the sputum sample will be sent to the Bacteriology, Virology and Mycology departments of CHRU Tours for characterization of microbial populations (Gram stain and bacterial cultures, Gomori-Grocott stain and fungal cultures, multiplex RTPCR for respiratory pathogens). The remaining sputum sample will then be sent to CEPR for pharmacological analyses of the IgG preparation. Unused or leftover samples will be kept at CEPR in a specific collection for further experimentation. They will be kept for an unrestricted period of time.

Blood samples will be sent to the Haematology and biochemistry laboratories for blood cell counts and C-Reactive Protein assays. 1 tube will be used for immunological analysis (neutrophil phenotyping, total IgG measurement) made at the CEPR.

No subject follow-up is scheduled as part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinical diagnosis of NCFB
* Computed tomography (CT) evidence of bilateral bronchiectasis
* Consent for research use of data and material
* Ability to provide an induced sputum sample
* Stable clinical status over the last 4 weeks

Exclusion Criteria:

* Pulmonary disease other than NCFB (except asthma)
* Diagnosis of cystic fibrosis
* Diagnosis of primary ciliary dyskinesia
* Requirement for oxygen therapy at rest
* Diagnosis of IgG deficiency (total serum IgG < 5.4 g/l)
* Treatment with a CFTR modulator drug in the last 6 months
* Unilateral bronchectasis
* CT evidence of interstitial lung disease with traction bronchectasis
* Refusal of the patient
* Acute exacerbation of NFCB in the last 4 weeks
* No sputum production
* Current treatment with systemic antibiotics (other than low dose azithromycin)
* Pregnancy or breastfeeding
* Subject under legal protection (e.g., guardianship, tutorship).
* Inability to produce a sputum sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Binding of Pseduomonas aeruginosa by a polyclonal IgG preparation in the presence of airway mucus obtained from patients with non-cystic fibrosis bronchiectasis | From enrollment to 3 months
  The main outcome is the quantification of polyclonal IgG binding to Pseudomonas aeruginosa in the presence of mucus derived from sputum of NCFB patients. Binding will be assessed by whole-cell ELISA.
  The results will be expressed as a percentage of binding over the one obtained when the polyclonal IgG is added in saline solution and will be compared with artificial mucus preparations in a range of viscosity similar to human airway mucus.

SECONDARY OUTCOMES:
Proteolysis of exogenous polyclonal IgG | From enrolment to 3 months
  The measurement of proteolysis, by Western-Blot, of exogenous polyclonal IgG added in the mucus derived from sputum of NCFB patients. The results will be expressed as a percentage of integrity over the one obtained when the polyclonal IgG is added in saline solution and will be compared with in vitro results.
Mobility of fluorescently labelled polyclonal IgG in mucus | From enrollment to 3 months
  The measurement of mobility by FRAP of exogenous fluorescently labelled polyclonal IgG added in the mucus derived from sputum of NCFB patients. The results will include the determination of the t(1/2), mobile and immobile fractions over the one obtained when the polyclonal IgG is added in saline solution and will be compared with in vitro results.
Impact of microbial airway colonization on IgG binding | From enrollment to 3 months
  Will be compared with uncolonized samples.
Impact of microbial airway colonization on proteolysis | From enrollement to 3 months
  Will be compared with uncolonized samples.
Impact of microbial airway colonization on Ig mobility | From enrollement to 3 months
  Will be compared with uncolonized samples.

OTHER OUTCOMES:
Comparaison between samples with microbial colonization (either bacterial, viral or fungal) and uncolonized samples. | From enrollement to 3 months
  Primary and secondary outcomes will be compared between samples with microbial colonization (either bacterial, viral or fungal) and uncolonized samples.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent PLANTIER, MD, Principal Investigator — CHRU de Tours
Locations (1):
- CHRU de Tours, Tours, France, France

IPD SHARING:
Plan to Share IPD: No